CLINICAL TRIAL: NCT03521752
Title: Influence of a Specific Exercise Program in the Institutionalized Elderly Balance
Brief Title: Influence of an Exercise Program in the Elderly Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Responsible Party: Principal Investigator, Cátia Filipa Flores Guimarães, Principal Investigator, Cooperativa de Ensino Superior, Politécnico e Universitário
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1CESPU
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Balance; Distorted
Keywords: BALANCE; INSTITUTIONALIZED ELDERLY PEOPLE; THERAPEUTIC EXERCISE; FUNCTIONAL CAPACITY

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Performed a specific program exercises (resistance training, balance, coordination and flexibility) during 4 weeks.
  Interventions: Other: Specific Exercise Program
- Control (No Intervention): The control group wasn't subjected to any intervention

INTERVENTIONS:
Other: Specific Exercise Program — 4 weeks of exercise classes, 2 to 3 times a week for a total of 10 sessions. Classes last approximately 40 minutes. The sessions included balance training, motor strength, endurance and flexibility. The training sessions were divided into warm-up, main activity and finally relaxation.
  Arms: Experimental

SUMMARY:
This study has the objective to determinate the effectiveness of a specific exercise program on balance and functional capacity of the daily activities of institutionalized elderly.

It was a randomized controlled trial with a total of 21 elderly that were randomly distributed into experimental (n = 11) and control groups (n=10). The experimental group performed a specific program exercises during 4 weeks, while the control group wasn't subjected to any intervention. Evaluations were carried out at the beginning and end of the exercise program, for both groups. After the intervention there were no statistically significant differences between groups in total balance and dynamic balance subscale, except static balance subscale.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* institutionalized elderly
* Both genders
* Mini-Mental ≥19 pontos
* Protocol attendance ≥ 90%

Exclusion Criteria:

* Cardiovascular diseases
* Contraindication to physical exercise
* Medication (anxiolytics, antidepressants)
* Vestibular disorders
* Previous physiotherapy of 6 months to the present study
* Neurological and neuromuscular diseases
* Use of gaiters
* Another type of physical exercise during the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-06-22 (Actual)

PRIMARY OUTCOMES:
Balance | 4 weeks
  Performance Oriented Mobility Assessment (POMA) This scale measures the static and dynamic balance, through the evaluation of some daily activities.
  This scale's scores are between 9 to 28 points, when 9 means hig risk of falling, and 28 means low risk of falling.
  It was used before and after the intervention.

SECONDARY OUTCOMES:
Functional capacity | 4 weeks
  Timed up and Go (TUG) This scale measures the mobility and locomotor performance, through the timing of an activity (lift from a chair, walk 3 meters, change direction and return to starting position).
  The cut-off points of the scale are divided into fully independent elderly (<10 seconds), independent elderly (10-19 seconds), and elderly people with difficulties in the tasks of daily living (20-29 seconds).
  It was evaluated before and after the intervention.